CLINICAL TRIAL: NCT02402920
Title: Phase I Trial of MK-3475 and Concurrent Chemo/Radiation for the Elimination of Small Cell Lung Cancer
Brief Title: Pembrolizumab and Concurrent Chemoradiotherapy or Radiation Therapy in Treating Patients With Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1003; NCI-2015-00598 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-1003 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-05

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma; Limited Stage Small Cell Lung Carcinoma; Neuroendocrine Neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (LS-SCLC, pembrolizumab, chemoradiotherapy) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and undergo radiation therapy BID 5 days a week for 3 weeks. Patients also receive cisplatin IV over 2 hours or carboplatin IV over 30 minutes and etoposide IV over 4 hours on days 1, 2, and 3. Treatment repeats every 3 weeks for 16 courses (1 course for radiation therapy, 4 courses for chemotherapy) in the absence of disease progression or unacceptable toxicity. Patients who achieve systemic disease control and do not exhibit severe (grade > 3) pembrolizumab related toxicity during/after completion of 16 courses may receive 16 additional courses of pembrolizumab in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Procedure: Radiation Therapy
- Part B (ES-SCLC, pembrolizumab, radiation therapy) (Experimental): Beginning after the completion of chemotherapy, patients receive pembrolizumab IV over 30 minutes on day 1 and undergo radiation therapy BID 5 days a week for 3 weeks. Treatment repeats every 3 weeks for 16 courses (1 course for radiation therapy) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Part A (LS-SCLC, pembrolizumab, chemoradiotherapy)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Part A (LS-SCLC, pembrolizumab, chemoradiotherapy)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
  Arms: Part A (LS-SCLC, pembrolizumab, chemoradiotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of pembrolizumab when given together with chemoradiotherapy or radiation therapy in treating patients with small cell lung cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving chemotherapy with radiation therapy may kill more cancer cells. Giving pembrolizumab with chemoradiotherapy or radiation therapy may be a better treatment for small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Safety of pembrolizumab (MK 3475) plus chemotherapy (chemo)/radiation for limited-stage small-cell lung cancer (LS-SCLC).

II. Safety of MK-3475 plus radiation for extensive-stage small-cell lung cancer (ES-SCLC).

SECONDARY OBJECTIVES:

I. MK-3475 will improve progression free survival (PFS) compared to historical controls for LS-SCLC and ES-SCLC.

OUTLINE: This is a dose-escalation study of pembrolizumab. Patients are assigned to either Part A or Part B based on diagnosis.

PART A (LS-SCLC): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and undergo radiation therapy twice daily (BID) 5 days a week for 3 weeks. Patients also receive cisplatin IV over 2 hours or carboplatin IV over 30 minutes and etoposide IV over 4 hours on days 1, 2, and 3. Treatment repeats every 3 weeks for 16 courses (1 course for radiation therapy, 4 courses for chemotherapy) in the absence of disease progression or unacceptable toxicity. Patients who achieve systemic disease control and do not exhibit severe (grade > 3) pembrolizumab related toxicity during/after completion of 16 courses may receive 16 additional courses of pembrolizumab in the absence of disease progression or unacceptable toxicity.

PART B (ES-SCLC): Beginning after the completion of chemotherapy, patients receive pembrolizumab IV over 30 minutes on day 1 and undergo radiation therapy BID 5 days a week for 3 weeks. Treatment repeats every 3 weeks for 16 courses (1 course for radiation therapy) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, all patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have a performance status of 0 or 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL (performed within 10 days of treatment initiation)
* Platelets >= 100,000/mcL (performed within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (performed within 10 days of treatment initiation)
* Serum creatinine or measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) or >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (creatinine clearance should be calculated per institutional standard) (performed within 10 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 X ULN or =< 5 X ULN for subjects with metastatic malignant neoplasm in the liver (liver metastases) (performed within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants, activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Histologic diagnosis of either limited stage SCLC (LS-SCLC), or extensive stage SCLC (ES-SCLC) or neuroendocrine tumor

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent (except glutamine) or using an investigational device within 2 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; with the exception of physiologic steroid replacement
* Has had a prior monoclonal antibody within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; prior radiation does not require a washout period; note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include skin basal cell carcinoma (basal cell carcinoma of the skin), skin squamous cell carcinoma (squamous cell carcinoma of the skin), or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed cell death-1 (PD-1), anti-programmed cell death-ligand 1 (PD-L1), anti-programmed cell death 1 ligand 2 (PD-L2), anti-cluster of differentiation (CD)137
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [HCV RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of pembrolizumab with concurrent chemoradiation determined by dose limiting toxicities graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Part A) | Up to 22 days after therapy initiation
  Frequency of adverse events will be tabulated by grade, type, and dose/cohort. Relative frequencies and confidence intervals will also be constructed.
Maximum tolerated dose of pembrolizumab with concurrent radiation determined by dose limiting toxicities graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Part B) | Up to 22 days after therapy initiation
  Frequency of adverse events will be tabulated by grade, type, and dose/cohort. Relative frequencies and confidence intervals will also be constructed.

SECONDARY OUTCOMES:
Response rate | Up to 8 years
  Will be performed using Global Immune Related Response Criteria that factors all indexed and non-indexed lesions, In-Field Immune Related Response Criteria in which only non-radiation therapy-treated lesions and non-index lesions arising outside the radiation therapy planning target volume will be considered, and Out-Field Immune Related Response Criteria in which only non-radiation therapy-treated lesions and non-index lesions arising outside the radiation therapy planning target volume will be considered.
Progression free survival | Up to 8 years
  Time to event distributions for progression free survival will be estimated via Kaplan-Meier analysis.
Overall survival | Up to 8 years
  Time to event distributions for overall response will be estimated via Kaplan-Meier analysis.
Biomarker response | Up to 8 years
  Descriptive analysis will include a global assessment of patient outcomes for parts A and B separately.

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Welsh JW, Heymach JV, Chen D, Verma V, Cushman TR, Hess KR, Shroff G, Tang C, Skoulidis F, Jeter M, Menon H, Nguyen QN, Chang JY, Altan M, Papadimitrakopoulou VA, Simon GR, Raju U, Byers L, Glisson B. Phase I Trial of Pembrolizumab and Radiation Therapy after Induction Chemotherapy for Extensive-Stage Small Cell Lung Cancer. J Thorac Oncol. 2020 Feb;15(2):266-273. doi: 10.1016/j.jtho.2019.10.001. Epub 2019 Oct 9. PMID 31605794
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org